CLINICAL TRIAL: NCT03702517
Title: Efficacy of Lateral Stair Walking Training in Patients With Chronic Stroke: a Pilot Randomized Controlled Study
Brief Title: Lateral Stair Walking Training After Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Wan-Yun Huang, Physical Therapist, Principal Investigator, Assistant Professor), Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VGHKS15-CT8-23
Record Dates: First submitted 2018-10-04; First posted 2018-10-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Chronic Stroke Patients
Keywords: lateral stair walking; range of motion; muscle strength
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lateral stair walking exercise (Experimental): The experimental group received 15 minutes of lateral stair walking exercise
  Interventions: Device: lateral stair walking exercise; Device: traditional physiotherapy
- traditional physiotherapy (Active Comparator): strengthening exercise, balance training and gait training
  Interventions: Device: lateral stair walking exercise; Device: traditional physiotherapy

INTERVENTIONS:
Device: lateral stair walking exercise — 15 minutes of lateral stair walking exercise
  Other Names: stair walking training
Device: traditional physiotherapy — strengthening exercise, balance training and gait training
  Other Names: physical therapy

SUMMARY:
The experimental group received 15 minutes of lateral stair walking exercise and 30 minutes of traditional physiotherapy (strengthening exercise, balance training and gait training) each time.

The measures were done by one experience physical therapist (not involve in the intervention) before receiving the intervention and at weeks four, eight, and twelve. It took 45 minutes for each subject to complete all measures each time.

DETAILED DESCRIPTION:
For lateral stair walking training, the dynamic stair trainer features four steps. The height can be adjusted from 0 to 16.5 centimeters, the stair was 0.74 m in width, with each step being 16 cm deep and 10 cm long. The experimental group received different heights of lateral stair walking training according to the patients' ability. The patients went up the stairs with the affected leg up first and they went down stairs with the sound leg leading first. For safety, the subjects held a handrail during the lateral stair walking exercise. The control group received traditional physiotherapy (strengthening exercise, balance training and gait training) for 30 minutes. Both the experimental group and control group received the intervention once a week for 12 weeks. All the interventions were done by the same physical therapist.

ELIGIBILITY:
Inclusion Criteria:

* subjects who were diagnosed with stroke within 6 months to 6 years by a neurologist or physiatrists,
* computerized tomography scan or magnetic resonance imaging scan showed unilateral brain damage,
* no obvious cognitive impairment,
* no serious bone and joint problems
* could follow the instructions and steps of the experiment
* walked 15 meters independently.

Exclusion Criteria:

* cognitively impaired,
* visually impairedor
* unable to receive training due to other diseases (lung, heart, gastrointestinal tract, bone and muscle, nervous system etc.)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01-03 (Actual); Primary Completion 2016-05-05 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
muscle strength | Both the experimental group and control group received the intervention once a week for 12 weeks.The measures were done by one experience physical therapist before receiving the intervention and at weeks four, eight, and twelve.
  Mycroft 3 hand-held dynamometer18: It has good reliability. Muscle strength can be measured in Newton's. It is applied in assessing the muscle strength of subjects.

SECONDARY OUTCOMES:
The postural assessment scale for stroke patients (PASS) | Both the experimental group and control group received the intervention once a week for 12 weeks.The measures were done by one experience physical therapist before receiving the intervention and at weeks four, eight, and twelve.
  The PASS assesses balance in lying, sitting and standing positions. It was designed specifically for patients with stroke and is suitable for all individuals regardless of postural performance. Its advantage lies in the lack of ceiling effect and floor effect, and the static and dynamic balance of stroke patients can be assessed. It is rated on a scale from 0 to 3, (total score of = 36) The Higher scores indicate better balance in stroke patients.
Fugal-Meyer assessment for Lower extremity, | Both the experimental group and control group received the intervention once a week for 12 weeks.The measures were done by one experience physical therapist before receiving the intervention and at weeks four, eight, and twelve.
  It is an assessment scale developed from Brunnstrom stage-L/E specifically dedicated to stroke patients. It is rated on a scale from 0 to 2. It has good reliability and validity.
Barthel index for Activities of Daily Living (ADL) | Both the experimental group and control group received the intervention once a week for 12 weeks.The measures were done by one experience physical therapist before receiving the intervention and at weeks four, eight, and twelve.
  It is a basic scale for functional independence with reliability and validity, covering 10 items such as eating, transposition, personal hygiene, using the bathroom, showering, walking on flat ground, stair climbing, putting on clothes, controlling excretion, etc. The total score ranges from 0 to 100, which is the progressive scope for activities of daily living .
Timed up and go test (TUG) | Both the experimental group and control group received the intervention once a week for 12 weeks.The measures were done by one experience physical therapist before receiving the intervention and at weeks four, eight, and twelve.
  In the Timed Up and Go Test time is recorded when rising from a chair, walking three metres, turning, and walking back. It has good sensitivity and specificity (sensitivity=87%, specificity=87%), and can assess balance and motor ability. The measured time can predict the fall of stroke patients.
Reha Gait® for gait parameters. | Both the experimental group and control group received the intervention once a week for 12 weeks.The measures were done by one experience physical therapist before receiving the intervention and at weeks four, eight, and twelve.
  It has high reliability. By wearing the three-axis gyro sensor on the shoes, gait data can be collected and analyzed with a microcomputer via Bluetooth.
Passive range of motion (PROM) | Both the experimental group and control group received the intervention once a week for 12 weeks.The measures were done by one experience physical therapist before receiving the intervention and at weeks four, eight, and twelve.
  Passive range of motion (PROM) and active range of motion (AROM) of hip, knee and ankle joints: The change in degree is measured with a goniometer before and after training.
active range of motion (AROM) | Both the experimental group and control group received the intervention once a week for 12 weeks.The measures were done by one experience physical therapist before receiving the intervention and at weeks four, eight, and twelve.
  Passive range of motion (PROM) and active range of motion (AROM) of hip, knee and ankle joints: The change in degree is measured with a goniometer before and after training.
The Brunnstrom motor recovery stage of Lower extremity (LE): | Both the experimental group and control group received the intervention once a week for 12 weeks.The measures were done by one experience physical therapist before receiving the intervention and at weeks four, eight, and twelve.
  The motor recovery was assessed using Brunnstrom motor recovery stage tool (Brunnstrom, 1970) that classifies it into 6 stages; 1) flaccidity; 2) spasticity is developing; 3) spasticity is maximum; 4) spasticity begins to decrease and some movement combinations become available; 5) spasticity is diminishing and more difficult movement combinations can be accomplish; 6) normal. It has good reliability and validity, and can assess the motor recovery of stroke patients. It is rated on a scale from 1 to 6.

CONTACTS AND LOCATIONS:
Overall Officials: I-Hsiu Liou, MD., Study Chair — Kaohsiung Veterans General Hospital.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Kaohsiung Veterans General Hospital — https://www.vghks.gov.tw/